CLINICAL TRIAL: NCT04975685
Title: Strengthening Mental Abilities With Relational Training (SMART) in Multiple Sclerosis (MS): A Feasibility Trial
Acronym: SMART_MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lincoln (Other)
Collaborators: University of Exeter (Other); Nottinghamshire Healthcare NHS Trust (Other Government); National University of Ireland, Maynooth (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21002
Record Dates: First submitted 2021-07-01; First posted 2021-07-23 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAU + SMART (Experimental): Participants in this arm will receive treatment-as-usual (TAU) plus the experimental SMART intervention (theory-based cognitive training)
  Interventions: Behavioral: SMART
- TAU + Sham training (Sham Comparator): Participants in this arm will receive treatment-as-usual (TAU) plus a control (sham) cognitive training intervention
  Interventions: Behavioral: Sham brain training (Sudoku)
- TAU (treatment-as-usual) (No Intervention): Participants in this arm will receive treatment-as-usual (TAU). Content of TAU for cognitive concerns, based on our clinical experience and knowledge, is often informational support from an MS Nurse with signposting to the MS Society/MS Trust websites.

INTERVENTIONS:
Behavioral: SMART — SMART (Strengthening Mental Abilities Through Relational Training) is a web-based cognitive training program that directly trains 'relational skills' - skills necessary to understand how concepts relate to one another, which underpin complex cognition.
  Arms: TAU + SMART
Behavioral: Sham brain training (Sudoku) — Sudoku was selected to control for expectancy effects based on popular conceptions that it broadly improves cognitive functions, coupled with little evidence supporting this notion, and its use as an active control in similar trials.
  Arms: TAU + Sham training

SUMMARY:
Background: Multiple Sclerosis (MS) is a chronic condition of the central nervous system; around 1 in 600 people in the United Kingdom have MS. Many people with MS (70%) have cognitive difficulties, which they experience as distressing and disabling, and there is currently a lack of treatment options to improve these difficulties.

SMART (Strengthening Mental Abilities with Relational Training) - a theory-based online cognitive training programme, which has been shown to improve general cognitive abilities - has not been tested with people who have MS.

Aims: To conduct a feasibility study to inform development of a definitive trial of SMART for improving cognitive functioning in people with MS. The investigators will assess:

1. Acceptability to participants of the intervention, delivery format, inclusion/exclusion criteria, baseline and outcome measures, randomisation protocol, and study procedures
2. The framework for a cost-effectiveness analysis alongside a definitive trial
3. Participant recruitment and retention rates
4. Sample-size needed for fully powered trial
5. Signal of efficacy

Plan: To address Aims 1-5, the investigators will recruit 60 adults with MS who are experiencing cognitive difficulties, identified from MS clinics.

Participants will complete baseline assessments of their cognitive abilities and answer questionnaires about their cognitive difficulties, personal priorities, mood, fatigue, self-efficacy, quality of life, and healthcare services used.

Assessments will be administered by a researcher, face-to-face or remotely.

Participants will be randomly allocated to one of three arms (20 per group):

Group 1: Receives SMART intervention online - plus usual care (MS Nurse support). SMART intervention involves completing a series of logic problems, which are designed to train skills that scaffold complex cognition.

Group 2: Receives usual care alone. Group 3: Receives a 'control' intervention online - plus usual care.

Baseline measures will be re-administered at three- and six-months post-randomisation. Researchers and patient-partners (people with personal experience of MS, who will act as co-researchers) will also interview 30 participants about their experience of the study and treatment. All qualitative data will be transcribed and thematically analysed in terms of a priori feasibility aims. Quantitative data will enable sample-size calculation for a definitive study and determine signal of efficacy.

DETAILED DESCRIPTION:
Background:

Cognitive deficits have been identified as the most debilitating impact of MS. These deficits interfere with daily living, manifesting as inattention (e.g., getting easily distracted), forgetting (e.g., leaving the stove on after cooking), and problem-solving difficulties (e.g., getting confused when completing a multi-stage task like cooking). The burden of these deficits reduces quality of life and restricts daily activities and employment - and correspondingly, diminishes patient perceptions of personal competence and self-worth. Cognitive rehabilitation is not routinely offered in the National Health Service (NHS) - and, when it is offered, largely focuses on teaching people to compensate for deficits (e.g., using external memory aids) rather than retraining cognitive skills. A recent state-of-the-field review from international MS experts has called for research towards identifying effective, evidence-based, and clinically feasible interventions to address cognitive deficits in MS. There is evident uncertainty about how to intervene effectively, and this is recognised by the James Lind Alliance as a top-10 priority area for research-funding.

Our trial tests the feasibility of a highly accessible and low-resource format of cognitive rehabilitation (online training). Given NHS resource constraints, the scale of the problem, and concerns about face-to-face consultation in the context of COVID-19, new and cost-effective ways of implementing promising cognitive rehabilitation interventions are needed. Low-resource online formats are more likely to be implemented if found to be clinically effective, enable wider access for patients, and provide active support for self-management - consistent with (1) models of care for managing longer-term conditions and (2) the digital healthcare agenda.

As a feasibility trial, outcomes are unlikely to immediately effect changes to NHS practice. However, this is a necessary step towards developing a definitive trial - and will give us a signal of efficacy, a prerequisite for progression to a definitive trial. If found to be clinically- and cost-effective, the latter trial could create a step-change in MS cognitive rehabilitation - improving service-delivery and optimising support with limited additional resources.

Aim:

To conduct a feasibility study to inform development of a definitive trial of SMART (an online 'brain training' treatment) for improving cognitive functioning in people with MS.

The investigators will assess:

1. Acceptability to participants of the intervention, delivery format, inclusion/exclusion criteria, baseline and outcome measures, randomisation protocol, and study procedures
2. The framework for a cost-effectiveness analysis alongside a definitive trial
3. Participant recruitment and retention rates
4. Sample-size needed for fully powered trial
5. Signal of efficacy

Research plan:

The investigators will conduct a three-arm feasibility Randomised Controlled Trial (RCT) comparing (1) SMART + treatment-as-usual (TAU) with (2) TAU and (3) active control ('sham') training + TAU.

Consenting eligible patients will complete a baseline cognitive assessment battery and questionnaires assessing impact of living with MS, health-related quality of life, subjective cognitive difficulties, and service/resource-use.

After completing baseline assessments, participants will be randomly allocated to one of three arms (using minimisation to balance participant characteristics across arms):

1. SMART + TAU
2. TAU. Content of TAU for cognitive concerns, based on our clinical experience and knowledge, is often informational support from an MS Nurse with signposting to the MS Society/MS Trust websites.
3. Sham training (active control: Sudoku) + TAU. The investigators selected Sudoku to control for expectancy effects based on popular conceptions that it broadly improves cognitive functions, coupled with little evidence supporting this notion, and its use as an active control in similar trials. Sham-training will be delivered online, over the same timeframe/regimen as SMART treatment, and with telephone support to facilitate access - controlling for modality, schedule of engagement, and relational support.

A Research Fellow will complete blinded outcomes at 3- and 6-months post-randomisation, by re-administering baseline measures. Quantitative data will enable sample-size calculation for a definitive study and determine signal of efficacy. After the first follow-up assessment (>3 months post-randomisation) a sub-sample of participants will engage in feasibility-feedback interviews.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS, received ≥3-months pre-enrolment (allowing for acute adjustment, as per other trials of cognitive rehabilitation)
* Age 18-89 (to meet the standardisation criteria of psychometric assessments)
* Cognitive difficulties as assessed by Perceived Deficits Questionnaire (PDQ) self-report (≥27) and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) testing (≤1 standard deviation below normative reference-value)
* Able to read and speak English to standard necessary for completing assessment and intervention procedures
* Able and willing to access a computer/tablet/smart-phone with internet connection throughout the study
* Able and willing to give informed consent

Exclusion Criteria:

* Currently receiving cognitive rehabilitation
* Previously received SMART training
* Vision or hearing problems precluding completion of procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rates | 16 months
  Numbers eligible/interested/consented and randomised (and reasons for non-participation), number completing baseline and outcome assessments at Follow-up 1
Completion rates of outcome measures | 6 months
  Missing response-data
Intervention drop-out rate | 3 months
  Numbers in the intervention condition that drop out (complete <6 sessions) and reasons for intervention non-completion

OTHER OUTCOMES:
Perceived Deficits Questionnaire (PDQ) | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
Symbol Digit Modalities Test (SDMT) | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
Generalized Anxiety Disorder Scale-7 (GAD-7) | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
Patient Health Questionnaire-9 (PHQ-9) | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
Modified Fatigue Impact Scale-5-Item (MFIS-5) | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
Personal Questionnaire (PQ) | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
EQ-5D-5L | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
MS Impact Scale-29 (MSIS-29) | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)
ICECAP-A | Change between baseline and 3-month follow-up. Additional follow-up at 6 months.
  Estimates of (group-level) effect-sizes with 95% Confidence Intervals (CIs) and proportions achieving reliable/clinically significant change (exploring signal of efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Nima Moghaddam, DClinPsy, Principal Investigator — University of Lincoln
Locations (1):
- Nottingham Centre for Multiple Sclerosis and Neuroinflammation, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Golijani-Moghaddam N, Dawson DL, Evangelou N, Turton J, Hawton A, Law GR, Roche B, Rowan E, Burge R, Frost AC, das Nair R. Strengthening Mental Abilities with Relational Training (SMART) in multiple sclerosis (MS): study protocol for a feasibility randomised controlled trial. Pilot Feasibility Stud. 2022 Sep 3;8(1):195. doi: 10.1186/s40814-022-01152-7. PMID 36056385